CLINICAL TRIAL: NCT03818321
Title: Methenamine Hippurate With Cranberry Capsules Versus Cranberry Capsules Alone for UTI Prevention in a Short-term Indwelling Foley Catheter Population After Urogynecological Surgery: A Double-Blinded Randomized Controlled Trial
Brief Title: Urinary Track Infection Prevention After Urogynecological Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18-115
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Urinary Tract Infections; Urinary Retention Postoperative; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Tract Infections; Pelvic Organ Prolapse | interventions — methenamine hippurate; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is randomized double-blinded placebo-controlled trial, and both patients and investigators are blinded. However, a research nurse will not be blinded to the group allocation, and the research nurse will order each patient's medication to the inpatient pharmacy based on the study randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methenamine Hippurate with Cranberry (Experimental): Subjects will be instructed to take Methenamine Hippurate 1 g tablet ( 1 tablet twice daily) with Cranberry supplementation (1 tablet twice daily) by mouth starting at time of discharge for 6-8 days.
  Interventions: Drug: Methenamine Hippurate 1 g tablet
- Placebo with Cranberry (Placebo Comparator): Subjects will be instructed to take Placebo tablet (1 tablet twice daily) with Cranberry supplementation (1 tablet twice daily) by mouth starting at time of discharge for 6-8 days.
  Cranberry capsules were incorporated into the standard practice of Cincinnati Urogynecology Associates, TriHealth Inc in mid-March 2016.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Methenamine Hippurate 1 g tablet — Methenamine Hippurate (study drug) is an FDA approved medication in the prevention of UTI. Methenamine Hippurate 1g contains Hippuric acid salt of Methenamine (hexamethylene tetramine), Magnesium Stearate, Povidone, Saccharin Sodium, FD&C Yellow No. 5 (tartrazine) (www.iodine.com/drug/hiprex/fda-package-insert).
  Arms: Methenamine Hippurate with Cranberry
Drug: Placebo tablet — Placebo is a tablet that will be provided to you that looks like the study drug but does not contain any medication. These pills are comprised of gelatin and minimal amounts of lactose powder. The pills are designed to have no effect on the patient.
  Arms: Placebo with Cranberry

SUMMARY:
This study is randomized double-blinded placebo-controlled trial to access oral Methenamine Hippurate (MH) in combination with cranberry capsules is superior to cranberry capsules alone in prevention of UTI in patients with transient post-operative urinary retention requiring a Foley catheter after pelvic reconstructive surgery.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are one of the most common bacterial infections in women. It is estimated that 1.6 billion dollars are spent on UTI treatment each year. Antibiotics have been the mainstay of treatment of UTIs, however frequent use has increased the prevalence of antibiotic resistant organisms. Therefore, focus has shifted to non-antibiotic therapy for UTI prophylaxis.

Methenamine Hippurate (MH) has been studied for decades due to its potential role in prevention of UTI. While not technically an antibiotic, MH works via its bacteriostatic action in the bladder. Benefits of MH are the lack of development of resistance, and the selective nature of this drug to the urinary system only. However, MH is best used in conjunction with an acidifying agent to increase its bioavailability (such as cranberry capsules or other acidic products). The usage of MH has been studied in various populations, has been seen to be effective in short-term catheterization. Usage of cranberry as prophylaxis for UTI is controversial; however, results have been favorable in the post-operative gynecological population.

Post-operative urinary retention (POUR) occurs frequently in patients who undergo incontinence and pelvic prolapse surgery. Although the definition of POUR can vary between clinicians, it is reported as 2.5-24% to as high as 43% after tension-free transvaginal mesh sling placement. This population is at also at high risk for UTI due to advanced age and menopausal status. Moreover, using a catheter longer than 2 days incurs a 2-fold increased risk of development of UTI with an estimated 5% increase in bacteriuria each day of catheterization.

In hopes to decrease the overuse of antibiotics and decrease the likelihood of antibiotic resistance, we propose that the use of MH and cranberry can reflect a potential benefit in this population of short-term indwelling Foley catheter use and help reduce the incidence of post-operative UTI after pelvic surgery.

The patients will then be randomized to either receive cranberry capsules and placebo OR cranberry capsules and Methenamine Hippurate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo major pelvic organ prolapse surgery that are diagnosed with POUR via failed retrograde void trial and require an indwelling Foley catheter upon hospital discharge.

Exclusion Criteria:

* Unwillingness to participate in the study
* Inability to understand English
* Pregnant women
* Patient personal history of nephrolithiasis, urogenital anomaly, neurogenic bladder, chronic renal insufficiency (GFR <60 ml/min/1.73 m² or serum creatinine level >1.03 for >3months), sarcoidosis, and severe hepatic insufficiency
* Currently (prior 3 months) undergoing medical management for recurrent UTI or interstitial cystitis
* Active urinary tract infection
* Patient history of taking Warfarin (Coumadin)
* Intraoperative bladder injury or cystotomy
* Physical or mental impairment that would affect the subject's ability to take medications daily or fill out questionnaires
* Reported allergy to any of the ingredients in the cranberry, MH, or placebo pill

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Tam TY, Aldrich ER, Crisp CC, Yook E, Yeung J, Pauls RN. Methenamine Hippurate With Cranberry Capsules Versus Cranberry Alone for Urinary Tract Infection Prevention in a Short-Term Indwelling Foley Catheter Population After Urogynecologic Surgery: A Double-Blinded Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2022 Mar 1;28(3):e55-e61. doi: 10.1097/SPV.0000000000001147. PMID 35272334

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo With Cranberry: Subjects will be instructed to take Placebo tablet (1 tablet twice daily) with Cranberry supplementation (1 tablet twice daily) by mouth starting at time of discharge for 6-8 days.
  Cranberry capsules were incorporated into the standard practice of Cincinnati Urogynecology Associates, TriHealth Inc in mid-March 2016.
  Placebo tablet: Placebo is a tablet that will be provided to you that looks like the study drug but does not contain any medication. These pills are comprised of gelatin and minimal amounts of lactose powder. The pills are designed to have no effect on the patient.
Period: Overall Study
Arm/Group | Methenamine Hippurate With Cranberry | Placebo With Cranberry
Started | 94 | 91
Completed | 93 | 89
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methenamine Hippurate With Cranberry | Placebo With Cranberry | Total
Number analyzed (Participants) | 93 | 89 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.27 (12.86) | 60.61 (12.44) | 60.95 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 89 | 182
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 85 | 85 | 170
  African American | 6 | 4 | 10
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 93 | 89 | 182

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Urinary Track Infection (UTI)
Description: Incidence of UTIs will be diagnosed at one week post-op visit.
Time Frame: From surgery to one week post-op visit, approximately 1 week post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Methenamine Hippurate With Cranberry | Placebo With Cranberry
Number analyzed (Participants) | 93 | 89
Participants | 62 | 71

ADVERSE EVENTS:
Time Frame: 6 week postop
Arm/Group | Methenamine Hippurate With Cranberry | Placebo With Cranberry
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/89
Other Adverse Events (participants affected / at risk) | 0/93 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT03818321/Prot_SAP_000.pdf